CLINICAL TRIAL: NCT05383755
Title: Development of a Digital Intervention to Address Stigma Among Pregnant Unmarried Adolescents Living With HIV
Brief Title: Digital Intervention to Address Stigma Among Pregnant Adolescents Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: Kenya Medical Research Institute (Other); 3-C Institute for Social Development (Industry); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Winfred K. Luseno, Senior Research Scientist, Pacific Institute for Research and Evaluation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R21TW011788 (NIH); 1805399 (Other: IRBNet); R21TW011788 (NIH)
Record Dates: First submitted 2022-05-12; First posted 2022-05-20 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Mother to Child Transmission; Pregnancy in Adolescence; Social Stigma; Self Disclosure; HIV
Keywords: HIV; Adolescent; Social Stigma; Mother-to-Child Transmission; Pregnancy in Adolescence; Software; Parents; Caregivers; Prevention; Self Disclosure; Cell Phone; Self Efficacy
MeSH Terms: conditions — Social Stigma | interventions — Seroconversion

STUDY DESIGN:
Intervention Model Description: The newly developed digital intervention uses illustrative characters to deliver didactic content to (1) raise awareness about stigma and its effects and understanding of disclosure and social support's importance, (2) increase self-efficacy and communication skills for disclosure and enlistment of caregivers as social support allies, and (3) tell stories to demonstrate how peers in similar situations have successfully coped with stigma, disclosed their pregnancies and/or HIV, and sought support from caregivers. Each module takes 20-30 minutes to complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital intervention (Experimental): Digital intervention for pregnant adolescents living with HIV.
  Interventions: Behavioral: Digital intervention for pregnant adolescents living with HIV

INTERVENTIONS:
Behavioral: Digital intervention for pregnant adolescents living with HIV — The newly developed digital intervention uses illustrative characters to deliver didactic content to (1) raise awareness about stigma and its effects and understanding of disclosure and social support's importance, (2) increase self-efficacy and communication skills for disclosure and enlistment of caregivers as social support allies, and (3) tell stories to demonstrate how peers in similar situations have successfully coped with stigma, disclosed their pregnancies and/or HIV, and sought support from caregivers. Each module takes 20-30 minutes to complete.

SUMMARY:
Pregnant adolescents living with HIV (ALHIV) in Kenya frequently experience stigma and difficulty telling a family member about their HIV and pregnancy status. This study will develop and evaluate a digital intervention for pregnant unmarried ALHIV to address the effects of stigma and strengthen communication skills. Family caregivers are an important yet underappreciated and understudied source of social support for pregnant unmarried ALHIV. The study will also identify acceptable approaches to involve family caregivers in addressing the detrimental effects of the intersecting stigmas faced by pregnant ALHIV. Together, these approaches are expected to improve engagement in PMTCT services among pregnant ALHIV. The study specific aims are to: (1) Develop and evaluate a digital intervention for pregnant unmarried ALHIV aged 15-19 to increase awareness of stigma and its consequences; improve disclosure self-efficacy and skills; and facilitate enlistment of family caregivers as social support allies to enhance uptake of PMTCT services; and (2) Identify acceptable approaches to increase awareness about stigma and enhance skills in communication and provision of social support among family caregivers. We will use data from individual interviews with pregnant ALHIV and joint interviews with pregnant ALHIV/caregiver dyads to develop initial intervention specifications and mock-ups. We will then conduct focus groups to obtain feedback on sample materials in order to refine the materials and develop an intervention prototype. We will then conduct a pilot to evaluate acceptability, usability, and preliminary efficacy of the prototype. All participating adolescents will receive a session in using the digital intervention with a mobile phone or tablet. The research team will ask questions both before the session and two weeks after the session in order to assess the intervention's usability and acceptability and preliminary improvements in the adolescents regarding stigma, disclosure, and social support. We will conduct focus groups with caregivers to identify acceptable approaches to involve them. Data will be used to finalize content and specifications of the digital intervention for pregnant ALHIV and will provide the framework for a future complementary intervention for caregivers, which will both be tested in a larger R34 or R01 trial.

DETAILED DESCRIPTION:
Our two-year study consisted of qualitative approaches for intervention development, and a single arm pre/post pilot study to assess the newly developed intervention's acceptability, usability, and preliminary efficacy (Aim 1). We also conducted focus group discussions (FGDs) with family caregivers to identify acceptable approaches to strengthen their supportive roles (Aim 2). For Aim 1, multi-methods were used spanning three phases: (1) in-depth interviews (IDIs) with pregnant adolescents living with HIV (ALHIV) and dyadic interviews (DIs) with ALHIV/caregiver pairs; (2) FGDs with ALHIV and (3) a pilot study with ALHIV. In the pilot study, we evaluated our newly developed digital intervention for pregnant adolescents living with HIV (ALHIV) in Kenya (N = 30). The intervention was designed to increase awareness of stigma regarding HIV and pregnancy, improve disclosure self-efficacy skills, and facilitate enlistment of family members as social support allies. The goal of the intervention was to enhance uptake of services for prevention of mother-to-child transmission of HIV (PMTCT). Using a single pre-post intervention group quasi-experimental design, the study assessed usability, acceptability, and preliminary improvements in stigma, disclosure, and social support measures. All participants received the intervention. The adolescents included in the pilot study were female, living with HIV, pregnant, unmarried, ages 15-19 years old. We included both rural and urban youth. There were two contacts with study participants. At the first contact, all participants were consented, completed a baseline quantitative survey, and received the intervention. During the intervention session, they were provided with a mobile phone/tablet with internet access, guided on how to access the digital intervention, received a guided tour of the website, and had their questions answered. After the tour, they were asked to review the intervention content. After reviewing the intervention content, participants completed a quantitative survey assessing the intervention's acceptability and usability. At the second contact, two weeks after the intervention session, follow up survey data was collected to assess maintenance/persistence of intervention effects after a short duration exposure. Survey measures at baseline and two-week follow up included demographics, stigma about HIV and pregnancy, disclosure self-efficacy for HIV and pregnancy, and disclosure of HIV and pregnancy to caregivers. Descriptive analyses were conducted of the quantitative data to describe time-related patterns and assess clinically meaningful improvements in our measures.

ELIGIBILITY:
Inclusion criteria for adolescent participants:

* Female
* Living with HIV
* Pregnant
* Unmarried
* 15-19 years old

Exclusion criteria for all participants:

* Does not meet all inclusion criteria
* Participated in a prior study activity
* Does not show adequate understanding of consent

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only female adolescents who are currently pregnant will be eligible to be in the study.
Enrollment: 169 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Winfred (Winnie) K. Luseno, PhD, Principal Investigator — Pacific Institute for Research and Evaluation
Locations (1):
- The Kenya Medical Research Institute - Centre for Global Health Research, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No
Because of the sensitive nature of the data and the small sample sizes, we are not planning to share the individual participant data in order to protect the confidentiality of study participants.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescents and caregivers were recruited with assistance from providers at health clinics.
Groups:
- Digital Intervention: Digital intervention for pregnant adolescents living with HIV: The digital intervention prototype sought to: (1) raise awareness about the intersecting stigmas of HIV and pregnancy; (2) strengthen self-efficacy and communication skills for disclosure and engagement of family caregivers as support allies; and (3) mitigate stigma's impact on disclosure and social support. We anticipated that these improvements would ultimately enhance PMTCT engagement and outcomes. The prototype was created in Adobe XD®, a software application used for designing and prototyping user interfaces (UI) and user experiences (UX) for web and mobile applications. The prototype was formatted for tablets and smart phones, used illustrative characters to engage, teach, and demonstrate key concepts, and featured limited interactivity that allowed users to click through using forward and back buttons.
Period: Aim 1 Phase 1: In-depth Interviews
Arm/Group | Digital Intervention
Started | 70 (Adolescents participated in either an individual in-depth interview (IDI; N=22) or a dyadic interview (DI) with their caregiver (N=24 adolescents and N=24 caregivers).)
Completed | 70
Not Completed | 0
Period: Aim 1 Phase 2: Adolescent Focus Groups
Arm/Group | Digital Intervention
Started | 22 (We conducted four focus group discussions (2 rural, 2 urban; n=22) to evaluate the intervention prototype and obtain feedback on intervention characteristics.)
Completed | 22
Not Completed | 0
Period: Aim 1 Phase 3: Pilot Clinical Trial
Arm/Group | Digital Intervention
Started | 30 (We conducted a pilot clinical trial single arm design to assess acceptability, usability, and preliminary efficacy of our digital intervention.)
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Aim 2 Round 1 Caregiver Focus Groups
Arm/Group | Digital Intervention
Started | 24 (We presented Aim 1 Phase 1 findings, obtained caregivers' perceptions about whether the findings resonated with their experiences, and explored acceptable approaches to involve caregivers in addressing stigma and disclosure faced by pregnant adolescents living with HIV.)
Completed | 24
Not Completed | 0
Period: Aim 2 Round 2 Caregiver Focus Groups
Arm/Group | Digital Intervention
Started | 23 (We presented the intervention prototype and asked for caregivers' views on the intervention, including acceptability of a complementary digital intervention for caregivers.)
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only Aim 1 Phase 3 pilot participants completed baseline, immediate post intervention, and two-week follow-up surveys. For analysis, we used data from 29 Aim 1 Phase 3 pilot participants.
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.9 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African (Kenyan) | 29
Internalized AIDS-Related Stigma Scale [Mean (Full Range); unit: scale score] — Measures internalized HIV-related stigma (or self-stigma) among people living with HIV/AIDS (e.g., "You feel guilty that you are HIV positive;" Response Options: Agree, Disagree).
  (4 summed items; scale score range 0-4 with higher values indicating more stigma; Baseline scale Cronbach alpha =.870)
  scale score | 1 [0 to 4]
HIV/AIDS Stigma Instrument - People Living with HIV (PWLA) [Mean (Full Range); unit: scale score] — Measures experienced stigma as perceived by people living with HIV (e.g., "Someone stopped being my friend;" Response Options: Never, Once or twice, Several times, Most of the time) (14 summed items; 4-pt scale 0-3; score range 0-42 with higher values indicating more stigma; Baseline Cronbach alpha = .919). Although 19 items were examined for the scale, we deleted variables with no variation in responses. We kept only the items that had variation at both time points.
  scale score | 2.59 [0 to 24]
Response to Stress Questionnaire - HIV/AIDS Stigma: Disengaging Coping Subscale [Mean (Full Range); unit: scale score] — Measures how much respondent uses avoidance, denial, and wishful thinking to cope with the stigma of HIV/AIDS (e.g. "I try not to think about the stigma of living with HIV. I try to forget all about it;" Response Options: Not at all, A little, Some, A lot).
  (4 summed items; 4-pt scale 1-4; score range 4-16 with higher values indicating poorer coping; Baseline Cronbach alpha = .958)
  scale score | 8 [4 to 16]
Internalized Pregnancy-Related Stigma Scale [Mean (Full Range); unit: scale score] — Adapted for pregnancy-related stigma from the Internalized AIDS-Related Stigma Scale. Measures internalized pregnancy-related stigma among adolescents (e.g., "You feel guilty that you are pregnant;" Response Options: Agree, Disagree) (4 summed items; scale score range 0-4 with higher values indicating more stigma; Baseline Cronbach alpha = .777)
  scale score | 1.34 [0 to 4]
Pregnancy-Related Experienced Stigma Scale [Mean (Full Range); unit: scale score] — Adapted from the HIV/AIDS Stigma Instrument - PWLA. Measures experienced stigma due to being pregnant. (e.g., "People sang offensive songs when I passed by;" Response Options: Never, Once or twice, Several times, Most of the time).
  (11 summed items; 4-pt scale 0-3; score range 0-33 with higher values indicating more stigma; Baseline Cronbach alpha = .850). Thirteen potential items were considered for the scale and 11 items remained after deleting those that lacked variation in responses.
  scale score | 2.14 [0 to 10]
Response to Stress Questionnaire - Pregnancy Stigma: Disengaging Coping Subscale [Mean (Full Range); unit: scale score] — Adapted from Response to Stress Questionnaire - HIV/AIDS Stigma: Disengaging Coping Subscale to measure how much respondent uses avoidance, denial, and wishful thinking to cope with pregnancy-related stigma (e.g., "I try not to think about the stigma of being pregnant. I try to forget all about it;" Response Options: Not at all, A little, Some, A lot).
  (4 summed items; 4-pt scale 1-4; score range 4-16 with higher values indicating poorer coping; Baseline Cronbach alpha = .876)
  scale score | 7.07 [4 to 16]
Self-efficacy to make an effective decision to disclose HIV status [Mean (Standard Deviation); unit: units on a scale] — Measures respondent's confidence in making an effective decision to disclose HIV status to a family member.
  Question Item: "How confident are you that you could make an effective decision of whether to tell a family member that you are HIV-positive?"
  (1 item; 11-pt scale: 0-10; 0=cannot do, 10=certain can do). Higher scores mean more confidence.
  units on a scale | 6.28 (4.0)
Self-efficacy for knowing it is safe to disclose HIV status [Mean (Standard Deviation); unit: units on a scale] — Measures respondent's confidence in knowing when it is safe to disclose HIV status to a family member.
  Question Item: "How confident are you that you could know whether it was safe to tell a family member parent that you are HIV-positive?"
  (1 item; 11-pt scale: 0-10; 0=cannot do, 10=certain can do). Higher scores mean more confidence.
  units on a scale | 6.24 (3.75)
Number of participants who report difficulty in disclosing HIV status [Count of Participants; unit: Participants] — Measures whether the respondent finds it difficult to disclose their HIV status to people.
  Question Item: "It is difficult to tell people about my HIV infection."
  (1 item; agree/disagree)
  Participants | 24
Self-efficacy to make an effective decision to disclose pregnancy [Mean (Standard Deviation); unit: units on a scale] — Adapted from self-efficacy to make an effective decision to disclose HIV status. Measures respondent's confidence in making an effective decision to disclose pregnancy to a family member.
  Question Item: "How confident are you that you could make an effective decision of whether to tell a family member that you are pregnant?"
  (1 item, 11-pt scale: 0-10; 0=cannot do, 10=certain can do). Higher scores mean more confidence.
  units on a scale | 5.10 (4.79)
Self-efficacy for knowing it is safe to disclose pregnancy [Mean (Standard Deviation); unit: units on a scale] — Adapted from self-efficacy in knowing when it is safe to disclose HIV status. Measures respondent's confidence in knowing when it is safe to disclose pregnancy to a family member.
  Question Item: "How confident are you that you could know whether it was safe to tell a family member parent that you are HIV-positive?
  (1 item, 11-pt scale: 0-10, 0=cannot do, 10=certain can do). Higher scores mean more confidence.
  units on a scale | 5.52 (4.76)
Number of participants who report difficulty in disclosing pregnancy [Count of Participants; unit: Participants] — Measures whether the respondent finds it difficult to disclose their pregnancy to people.
  Question Item: "It is difficult to tell people about my HIV infection."
  (1 item; agree/disagree)
  Participants | 22
Family social support [Mean (Full Range); unit: scale score] — Measures how much support the respondent feels she has in her life from her family.
  Example item: "Family will always be there for me" (5-pt response scale of 0="Not at all like me" to 4="Very much like me").
  (6 summed items; score range 0-24 with higher values indicating greater support; Baseline Cronbach alpha = .866)
  scale score | 17.31 [1 to 24]
Medical Outcomes Study (MOS) Social Support [Mean (Full Range); unit: scale score] — Measures multiple dimensions of support, including emotional, informational, tangible, affectionate, and positive social interaction.
  Example item: "Someone you can count on to listen to you when you need to talk." (5-point response scale of 0="None of the Time" to 4="All of the Time").
  (19 summed items; score range 0-76 with higher values indicating greater support; Baseline Cronbach alpha = .937)
  scale score | 54.41 [24 to 76]
Center for Epidemiologic Studies Depression Scale Short Form 10 (CES-D 10) [Mean (Full Range); unit: scale score] — Measures depressive symptoms among general and clinical populations in the past 7 days. Example item: "How often did you feel that you could not 'get going'? (4-pt scale of 0="Rarely (<1 day) to 3="Most or all of the time (5-7 days)".
  (10 summed items; score range 0-30 with higher values indicating more depression symptomology; Baseline Cronbach alpha = .814)
  scale score | 7.52 [0 to 25]
Generalized Anxiety Disorder Scale 7 Items (GAD 7) [Mean (Full Range); unit: scale score] — Used for screening for generalized anxiety symptomology and assessing severity over last two weeks in clinical practice and research.
  Example item: "How often have you felt nervous, anxious or on edge" (4-pt response scale of 0="Rarely" (<1 day) to 3="Most or all of the time (5-7 days)".
  (7 summed items; score range 0-21 with higher values indicating more anxiety symptomology; Baseline Cronbach alpha = .871)
  scale score | 5.03 [0 to 17]

OUTCOME MEASURES:

1. Primary Outcome: User Version Mobile Application Rating Scale (uMARS) - Objective Quality Measure
Description: Aim 1 Phase 3 Acceptability of Final Prototype. Quantitative measure adapted for this study; overall objective quality (engagement, functionality, aesthetics, information); self-report survey items assessing overall objective quality of the digital intervention. Scale title: Adapted User version Mobile Application Rating Scale (uMARS; Low quality=1, High quality =5). App objective quality mean scores Min=4.25, Max=5.00. Higher scores mean perception of higher quality.
Time Frame: Immediately post-intervention approximately 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
score on a scale | 4.81 (0.22)

2. Primary Outcome: User Version Mobile Application Rating Scale (uMARS) - Subjective Quality Measure (Composite Measure)
Description: Aim 1 Phase 3 Acceptability of Final Prototype. Quantitative data; overall subjective quality; self-report survey items assessing overall subjective quality of the digital intervention. Scale title: Adapted User version Mobile Application Rating Scale (uMARS; Low quality=1, High quality =5). App subjective quality mean scores: Min=3.67, Max=5.00. Higher scores indicate perception of higher quality.
Time Frame: Immediately post-intervention approximately 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
score on a scale | 4.67 (0.47)

3. Primary Outcome: HIV/AIDS Stigma Instrument - People Living With HIV (PWLA)
Description: Aim 1 Phase 3. Change in perception of experienced stigma (e.g., "Someone stopped being my friend.") (Never, Once or twice, Several times, Most of the time)(14 summed items; scale score range 0-42 with higher values indicating more stigma)
Time Frame: Two weeks post-intervention
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
score on a scale | 2.31 [0 to 28]
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = -0.28 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

4. Primary Outcome: Internalized Pregnancy-Related Stigma Scale
Description: Aim 1 Phase 3. Change in internalized pregnancy-related stigma among adolescents. Example item:"Becoming pregnant and having a baby as a teen makes me feel ashamed and bad about myself;" Response Options: Agree, Disagree) (4 summed items; scale score range 0-4 with higher values indicating more stigma).
  Adapted for pregnancy-related stigma from the Internalized AIDS-Related Stigma Scale.
Time Frame: Two weeks post-intervention
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
score on a scale | 1 [0 to 4]
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = -0.34 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

5. Primary Outcome: Self-efficacy to Make an Effective Decision to Disclose HIV Status
Description: Aim 1 Phase 3. Change in the respondent's confidence in making an effective decision to disclose HIV status to a family member.
  Question Item: "How confident are you that you could make an effective decision of whether to tell a family member that you are HIV-positive?"
  (1 item; 11-pt scale: 0-10; 0=cannot do, 10=certain can do). Higher scores mean more confidence.
Time Frame: Two weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
units on a scale | 7.66 (3.59)
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = 1.38 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

6. Primary Outcome: Self-efficacy to Make an Effective Decision to Disclose Pregnancy
Description: Aim 1 Phase 3. Change in respondent's confidence in making an effective decision to disclose pregnancy to a family member.
  Question Item: "How confident are you that you could make an effective decision of whether to tell a family member that you are pregnant?"
  (1 item, 11-pt scale: 0-10; 0=cannot do, 10=certain can do; higher scores mean higher confidence).
  Adapted from self-efficacy to make an effective decision to disclose HIV status.
Time Frame: Two weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
units on a scale | 8.14 (3.81)
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = 3.03 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

7. Secondary Outcome: Self-efficacy for Knowing it is Safe to Disclose HIV Status
Description: Measures respondent's confidence in knowing when it is safe to disclose HIV status to a family member.
  Question Item: "How confident are you that you could know whether it was safe to tell a family member parent that you are HIV-positive?"
  (1 item; 11-pt scale: 0-10; 0=cannot do, 10=certain can do). Higher scores mean more confidence.
Time Frame: Two weeks post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
units on a scale | 7.59 (3.79)
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = 1.35 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

8. Secondary Outcome: Internalized AIDS-Related Stigma Scale
Description: Change in internalized HIV-related stigma (or self-stigma) among adolescents (e.g., "You feel guilty that you are HIV positive;" Response Options: Agree, Disagree).
  (4 summed items; scale score range 0-4 with higher values indicating more stigma)
Time Frame: Two weeks post-intervention
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
score on a scale | .55 [0 to 4]
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = -0.45 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

9. Secondary Outcome: Response to Stress Questionnaire - HIV/AIDS Stigma: Disengaging Coping Subscale
Description: Change in respondent's use of avoidance, denial, and wishful thinking to cope with the stigma of HIV/AIDS (e.g. "I try not to think about the stigma of living with HIV. I try to forget all about it;" Response Options: Not at all, A little, Some, A lot).
  (4 summed items; score range 4-16 with higher values indicating poorer coping)
Time Frame: Two weeks post-intervention
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 29
score on a scale | 6.66 [4 to 16]
Statistical Analysis 1: Comparison: Digital Intervention; Test type: Other — Single group; Mean Difference (Net) = -1.35 — Estimated value is the mean change value calculated between baseline and two weeks post-intervention

10. Secondary Outcome: Qualitative Theme, Disclosure Experiences. Sub-Theme: Direct Disclosure
Description: Data were collected for Aim 1 Phase 1. Measure Definition: Adolescent directly informs her caregiver that she is pregnant and/or living with HIV.
Time Frame: Single interviews were done during Aim 1 Phase 1 over a 4-month period (April - July 2022). Each interview lasted about 1 hour.
Population: The total number of participants in Aim 1 Phase 1 IDIs and DIs was 70, which included 46 adolescents and 24 caregivers. However, we used n=46 adolescents as our denominator or number analyzed because the focus of this phase was adolescents experiences.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants | 11

11. Secondary Outcome: Qualitative Theme, Disclosure Experiences. Sub-Theme: Indirect Disclosure
Description: Data were collected for Aim 1 Phase 1. Measure Definition: Adolescent makes no direct effort to reveal her status.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants | 2

12. Secondary Outcome: Qualitative Theme, Disclosure Experiences. Sub-Theme: Caregiver Initiated Disclosure
Description: Data were collected for Aim 1 Phase 1. Measure Definition: Caregiver informs the adolescent or otherwise initiates a discussion that reveals the status.
Time Frame: as for outcome 10
Population: The total number of participants in Aim 1 Phase 1 IDIs and DIs was 70, which included 46 adolescents and 24 caregivers. We used N=46 adolescents as our denominator or number analyzed because the focus of this phase was adolescents experiences.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants | 20

13. Secondary Outcome: Qualitative Theme, Disclosure Experiences. Sub-Theme: Mediated Disclosure
Description: as for outcome 12
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants | 18

14. Secondary Outcome: Qualitative Theme, Disclosure Experiences. Sub-Theme: Accidental Disclosure
Description: Data were collected during Aim 1 Phase 1. Measure Definition: The disclosure occurs though it was unintended by the adolescent.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants | 5

15. Secondary Outcome: Qualitative Theme, Perceptions About Stigma. Sub-Theme: HIV-Related Stigma Worse Than Pregnancy-Related Stigma
Description: Data were collected during Aim 1 Phase 1. Measure Definition: Adolescents who made statements suggesting that HIV-related stigma is worse than stigma associated with pregnancy.
Time Frame: as for outcome 10
Population: The total number of participants in Aim 1 Phase 1 IDIs and DIs was 70, which included 46 adolescents and 24 caregivers. However, we used n=46 adolescents as our denominator or number analyzed because the focus of this phase was adolescents experiences. HIV versus pregnancy-related stigma was not discussed with adolescents in 19 interviews. Thus, 27 participants were evaluated for this theme.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 27
Participants | 19

16. Secondary Outcome: Qualitative Theme, Perceptions About Stigma. Sub-Theme: Pregnancy-Related Stigma is Worse Than HIV-Related Stigma
Description: Data were collected during Aim 1 Phase 1. Measure Definition: Adolescents who made statements suggesting that pregnancy-related stigma is worse than stigma associated with HIV.
Time Frame: as for outcome 10
Population: The total number of participants in Aim 1 Phase 1 IDIs and DIs was 70, which included 46 adolescents and 24 caregivers. We used N=46 adolescents as our denominator or number analyzed because the focus of this phase was adolescents experiences. HIV versus pregnancy-related stigma was not discussed with adolescents in 19 interviews. Thus, 27 participants were evaluated for this theme.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 27
Participants | 6

17. Secondary Outcome: Qualitative Theme, Perspectives About Stigma. Sub-Theme: HIV-Related and Pregnancy-Related Stigma Equally Bad
Description: Data were collected during Aim 1 Phase 1. Measure Definition: Adolescents who made statements suggesting that HIV- and pregnancy-related stigma are equally bad.
Time Frame: as for outcome 10
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 27
Participants | 2

18. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: No Support Received
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who noted having not received support (e.g., money, food, clothing, encouragement, emotional support, etc.) that they needed.
Time Frame: as for outcome 10
Population: The total number of participants in Aim 1 Phase 1 IDIs and DIs was 70, which included 46 adolescents and 24 caregivers. We used N=46 adolescents as our denominator or number analyzed because the focus of this phase was adolescents experiences. Social support received before versus after disclosure of status was not discussed with adolescents in eight interviews. Thus, 38 participants were evaluated for this theme.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 22

19. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: Support Improved After Pregnancy Disclosure
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who thought the social support they received improved after disclosing their pregnancies.
Time Frame: as for outcome 10
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 5

20. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: Support Worsened After Pregnancy Disclosure
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who thought the social support they received worsened after disclosing their pregnancies.
Time Frame: as for outcome 10
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 12

21. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: Support Improved After HIV Disclosure
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who thought the social support they received improved after disclosing HIV.
Time Frame: as for outcome 10
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 0

22. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: Support Worsened After HIV Disclosure
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who thought the social support they received worsened after disclosing HIV.
Time Frame: as for outcome 10
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 2

23. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: No Change in Support After Pregnancy Disclosure
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who reported no change regarding the social support they received after having disclosed their pregnancy.
Time Frame: as for outcome 10
Population: The total number of participants in Aim 1 Phase 1 IDIs and DIs was 70, which included 46 adolescents and 24 caregivers. We used N=46 adolescents as our denominator or number analyzed because the focus of this phase was adolescents experiences. Social support received before versus after disclosure of status was not discussed with adolescents in eight interviews. Thus, 38 participants contributed to analysis of this theme.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 19

24. Secondary Outcome: Qualitative Theme, Perceptions About Social Support. Sub-Theme: No Change in Support After HIV Disclosure
Description: Data were collected during Aim 1 Phase 1. Responses from adolescents concerning their experiences and thoughts about social support received before and after their disclosure of HIV and/or pregnancy. Measure Definition: Adolescents who reported no change regarding the social support they received after having disclosed HIV.
Time Frame: as for outcome 10
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 38
Participants | 4

25. Secondary Outcome: Qualitative Theme: Number of Adolescents Who Reported That Their Caregivers Were Aware About Their Pregnancy at Time of Their Interview.
Description: Data were collected for Aim 1 Phase 1. Measure Definition: Adolescents reported whether, at the time of the interview, their primary caregiver knew about their pregnancy.
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants
  Caregiver knew about adolescent's pregnancy | 44
  Caregiver did not know about pregnancy | 2

26. Secondary Outcome: Qualitative Theme: Number of Adolescents Who Reported That Their Caregivers Were Aware About Their HIV Status at Time of Their Interview.
Description: Data were collected for Aim 1 Phase 1. Measure Definition: Adolescents reported whether, at the time of their interview, their primary caregiver knew about their HIV status.
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 46
Participants
  Caregivers were aware of adolescent's HIV status because they were diagnosed in early life | 32
  Caregivers were aware of adolescent's HIV status because adolescent disclosed their status | 12
  Caregivers were not aware about adolescent's HIV status because adolescent had not disclosed | 2

27. Secondary Outcome: Acceptability of Initial Prototype: Colors Used
Description: Data were collected for Aim 1 Phase 2. Four focus groups conducted with N=22 adolescents in total. Participants began by individually reviewing the initial prototype using a tablet and then used a rating form to share their perspectives about various features of the prototype. Intervention features rated by participants included color scheme, characters, backgrounds, story, and message. The rating form provided a star ranking system ranging from 1 (terrible) to 5 (excellent). The rating form was created specifically for this study.
Time Frame: Focus groups for Aim 1 Phase 2 were done over a 2-month period (May - June 2023). Participants took part in one focus group. Focus groups lasted on average 1 hour and 40 minutes.
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.45 (0.80)

28. Secondary Outcome: Acceptability of Initial Prototype: Adolescent Character
Description: Data collected for Aim 1, Phase 2. Four focus groups conducted with N=22 adolescents in total. Participants began by individually reviewing the initial prototype using a tablet and then used a rating form to share their perspectives about various features of the prototype. Intervention features rated by participants included color scheme, characters, backgrounds, story, and message. The rating form provided a star ranking system ranging from 1 (terrible) to 5 (excellent). The rating form was created specifically for this study.
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.23 (0.97)

29. Secondary Outcome: Acceptability of Initial Prototype: Healthcare Provider Character
Description: Data collected for Aim 1 Phase 2. Four focus groups conducted with N=22 adolescents in total. Participants began by individually reviewing the initial prototype using a tablet and then used a rating form to share their perspectives about various features of the prototype. Intervention features rated by participants included color scheme, characters, backgrounds, story, and message. The rating form provided a star ranking system ranging from 1 (terrible) to 5 (excellent). The rating form was created specifically for this study.
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.86 (0.47)

30. Secondary Outcome: Acceptability of Initial Prototype: Sister Character
Description: as for outcome 29
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.23 (0.97)

31. Secondary Outcome: Acceptability of Initial Prototype: Mother Character
Description: as for outcome 29
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.14 (0.83)

32. Secondary Outcome: Acceptability of Initial Prototype: Father Character
Description: as for outcome 29
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 3.77 (0.92)

33. Secondary Outcome: Acceptability of Initial Prototype: Brother Character
Description: as for outcome 29
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 3.50 (1.06)

34. Secondary Outcome: Acceptability of Initial Prototype: Home Background
Description: as for outcome 29
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.67 (0.58)

35. Secondary Outcome: Acceptability of Initial Prototype: Health Facility Background
Description: as for outcome 27
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.68 (0.65)

36. Secondary Outcome: Acceptability of Initial Prototype: Story
Description: as for outcome 27
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.73 (0.55)

37. Secondary Outcome: Acceptability of Initial Prototype: Message
Description: as for outcome 27
Time Frame: as for outcome 27
Population: A total of 22 pregnant adolescents participated in Aim 1 Phase 2 focus groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Digital Intervention
Number analyzed (Participants) | 22
score on a scale | 4.82 (0.39)

38. Secondary Outcome: Qualitative Theme, Caregivers' Perceptions About Engaging Them: Liked Idea of App for Caregivers
Description: Data were collected during Aim 2 Rounds 1 and 2. Frequencies of responses from caregivers concerning the intervention prototype and a potential complementary digital intervention for caregivers from four focus groups which included a total of 47 caregivers. Measure Definition: Caregivers who liked the idea of developing a similar digital intervention (i.e., an "App") for caregivers.
Time Frame: Focus groups were done during Aim 2 Rounds 1 and 2 in June and December 2023. Caregivers took part in one focus group. Each focus group lasted 2 hours.
Population: The total number of participants in Aim 2 focus groups was 47 caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 47
Participants | 16

39. Secondary Outcome: Qualitative Theme, Caregivers' Perceptions About Engaging Them: Preferred Engagement in Group Setting
Description: Data were collected during Aim 2 Rounds 1 and 2. Frequencies of responses from caregivers concerning the intervention prototype and a potential complementary digital intervention for caregivers from four focus groups which included a total of 47 caregivers. Measure Definition: Caregivers who preferred to be engaged in a group setting as an alternative to using an App.
Time Frame: as for outcome 38
Population: The total number of participants in Aim 2 focus groups was 47 caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 47
Participants | 5

40. Secondary Outcome: Qualitative Theme, Caregivers' Perceptions About Engaging Them: Preferred Engagement Via Written Media
Description: Data were collected for Aim 2 Rounds 1 and 2. Frequencies of responses from caregivers concerning the intervention prototype and a potential complementary digital intervention for caregivers from four focus groups which included a total of 47 caregivers. Measure Definition: Caregivers who preferred to be engaged in a group setting as an alternative to using an App.
Time Frame: as for outcome 38
Population: The total number of participants in Aim 2 focus groups was 47 caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 47
Participants | 4

41. Secondary Outcome: Qualitative Theme, Caregivers' Perceptions About Engaging Them: Preferred Engagement Via Radio Advertisements.
Description: Data were collected for Aim 2 Rounds 1 and 2. Frequencies of responses from caregivers concerning the intervention prototype and a potential complementary digital intervention for caregivers from four focus groups which included a total of 47 caregivers. Measure Definition: Caregivers who preferred to be engaged via radio advertisements as an alternative to using an App.
Time Frame: as for outcome 38
Population: The total number of participants in Aim 2 focus groups was 47 caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 47
Participants | 1

42. Secondary Outcome: Qualitative Theme, Caregivers' Perceptions About Engaging Them: Preferred Engagement in Healthcare Setting.
Description: Data were collected for Aim 2 Rounds 1 and 2. Frequencies of responses from caregivers concerning the intervention prototype and a potential complementary digital intervention for caregivers from four focus groups which included a total of 47 caregivers. Measure Definition: Caregivers who preferred to be engaged in a healthcare setting as an alternative to using an App.
Time Frame: as for outcome 38
Population: The total number of participants in Aim 2 focus groups was 47 caregivers.
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Intervention
Number analyzed (Participants) | 47
Participants | 1

ADVERSE EVENTS:
Time Frame: Individuals took part in five different research activities. An individual could only take part in one activity. Adverse event data were monitored as follows: Aim 1 Phase 1 - from enrollment to end of interview, about 1 week. Aim 1 Phase 2 - from enrollment to end of focus group, about 2 weeks . Aim 1 Phase 3 - (Pilot trial) from enrollment to end of follow-up, about 3 weeks. Aim 2 Rounds 1 and 2 - from enrollment to end of the focus group, about 2 weeks.
Groups:
- Digital Intervention: Digital intervention for pregnant adolescents living with HIV.
  Digital intervention for pregnant adolescents living with HIV: The newly developed digital intervention will include SMS for reminder purposes and Web-based components such as virtual simulations and didactic content to educate and build relevant skills (e.g., disclosure self-efficacy) to facilitate social support from caregiving family members. The intervention will (1) raise awareness about the intersecting stigmas of HIV and pregnancy; (2) highlight the effects of these stigmas on disclosure and social support; and (3) increase self-efficacy and communication skills for disclosure and enlistment of family members as social support allies. The goal of the intervention is to improve PMTCT engagement among pregnant unmarried ALHIV. Our theory-informed Web-based intervention will be use 3C Institute's Dynamic e-Learning Platform (DeLP), a customizable software platform that implements the evidence-based cognitive theory of multimedia learning (CTML) to effectively engage users.
Arm/Group | Digital Intervention
All-Cause Mortality (participants affected / at risk) | 0/169
Serious Adverse Events (participants affected / at risk) | 0/169
Other Adverse Events (participants affected / at risk) | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT05383755/Prot_SAP_000.pdf